CLINICAL TRIAL: NCT06443229
Title: Effect of Telerehabilitation Use in the Treatment of Non-specific Chronic Low Back Pain in the Brazilian Afrodescendants Population: a Randomized Controlled Trial Protocol
Brief Title: Effect of Telerehabilitation Use in the Treatment of Non-specific Chronic Low Back Pain in the Brazilian Afrodescendants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5.991.168
Record Dates: First submitted 2024-05-14; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-03

CONDITIONS: Telerehabilitation; Low Back Pain
Keywords: Telerehabilitation; Low Back Pain; Black People; Pain; Disability; Rehabilitation; Health of Ethnic Minorities
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized controlled double-blind clinical trial, with a 1:1 allocation of 102 participants divided into two groups (intervention or control).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be evaluated pre- and post-intervention by a blind evaluator, previously trained to obtain information and confirm eligibility criteria, in addition to primary and secondary outcomes. The evaluator will be asked to guess which group the participants were in (intervention or control) at the end of the study to measure the blindness of the evaluator. Regarding the data analyst, he will be blind to carry out this stage of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Activity based in exercises and educational approach (Experimental): Exercises for warming up, strengthening, and relaxation, along with informational sessions incorporating an educational approach for low back pain using Telerehabilitation platform.
  Interventions: Behavioral: Graded Activity based in exercises and educational approach
- Educational Approach (Sham Comparator): Educational approach for low back pain using Telerehabilitation platform.
  Interventions: Other: Educational Approach

INTERVENTIONS:
Behavioral: Graded Activity based in exercises and educational approach — Exercises for warming up, strengthening, and relaxation, along with informational sessions incorporating an educational approach for low back pain using Telerehabilitation platform. Participants will be randomized into two groups: the Experimental Group (EG), which will receive graded activity along with the educational approach, three times a week, over 12 sessions, totaling 4 weeks.
  The intervention will involve adapting a protocol from an exercise program based on gradual activity with progressively increasing exercise intensity using web applications from Physitrack® Ltd., LDN, United Kingdom (used by the physiotherapist/researcher) and Physiapp® (used by the participant). Participants will be provided with (i) a welcome letter outlining the intervention/group components they are allocated to; (ii) instructions on how to use the Physiapp® web application (web browser, Android or iOS app) at home.
  Arms: Graded Activity based in exercises and educational approach
Other: Educational Approach — Educational approach for low back pain using Telerehabilitation platform. Participants will receive educational materials with an isolated educational approach, with the delivery of the materials occurring three times a week.
  Arms: Educational Approach

SUMMARY:
The goal of this study is to measure the effect of telerehabilitation on the treatment of nonspecific chronic LBP in the adults Brazilian Black population. The main questions it aims to answer are:

1. Will the graded activity exercises guided by educational approach or only the educational approach alone improve low back pain intensity, functional capacity, quality of life, anxiety, fear-avoidance beliefs due to nonspecific chronic low back pain before, immediately after the 4-week intervention, and after 3 and 6 months of follow-up?
2. How will participants' behaviors in terms of frequency and adherence, exercise feedback diary, and educational approach for nonspecific chronic low back pain be?

   What are the participants' opinions and any difficulties or barriers encountered throughout the study?
3. What are the perceptions of discrimination based on race, gender, age, socioeconomic status, and education when accessing healthcare services for the treatment of low back pain in the past?

Researchers will compare Group Experimental Graded Activity with Educational Program with Telerehabilitation to a placebo (only Educational Approach ) to see improve the pain intensity and functional capacity because of low back pain.

Participants will:

* Take Group Experimental (GAEP) or a placebo (OEA) 3 times per week, for 1 month.
* Keep a feedback diary of their symptoms and the barriers they have.
* Visit the researcher by online teleassessment after one month, 3 months and 6 months follow-up.

DETAILED DESCRIPTION:
Background: Low back pain (LBP) is highly prevalent, ranging from 30 to 70% in developed and industrialized countries, leading to health costs and work absenteeism. However, when it comes to the Black population, studies addressing the treatment of nonspecific chronic LBP while considering the specificities of this population are scarce. The use of telerehabilitation opens up opportunities for the physiotherapy community to address musculoskeletal conditions.

The goal of this study is to measure the effect of telerehabilitation on the treatment of nonspecific chronic LBP in the adult Brazilian Black population.

Methods: A randomized controlled double-blind clinical trial, with a 1:1 allocation of 102 Afro-Brazilian participants divided into two groups, with 51 participants in each, experiencing nonspecific chronic LBP for at least 3 months, of both sexes, aged 18-65 years, residing in Brazil, and divided into the Gradual Activity Group (GAG) and Control Group (CG), with a duration of 12 sessions, three times per week. The intervention will involve the adaptation of an exercise program protocol based on gradual activity with progressive exercise intensity, through the web applications Physitrack® (researcher) and Physiapp® (participant). Sociodemographic and clinical characteristics will be evaluated. The primary outcome will be pain intensity, and secondary outcomes will include functional capacity, quality of life, beliefs, and fears. Also the perceptions of discrimination based on race, gender, age, socioeconomic status, and education will be assessed regarding prior access to healthcare services for the treatment of LBP. The groups will be assessed at baseline (T0), immediately post-treatment (T1), at 3-months (T2) and 6-months (T3) follow-ups. Data will be collected and managed using the REDCap® electronic data capture tools.

Discussion: Evidence suggests that telerehabilitation can be utilized as a potential tool to promote the treatment of non-severe conditions of nonspecific chronic LBP, but few studies have investigated the Black population while considering the specificities of populations that historically suffer from social inequalities in accessing healthcare treatments.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black (Black or Brown), according to Brazilian Institute of Geography and Statistics (IBGE) classification;
* Age range from 18 to 65 years old;
* Both biological sexes (female and male);
* Sedentary or physically active participants;
* Present chronic low back pain with a score ≥ 3 on the Numeric Pain Rating Scale for more than 3 months and due to nonspecific causes;
* Able to read, write, and speak Brazilian Portuguese;
* Live in Brazil in urban or rural areas;
* Have access to the internet;
* Possess a device with internet access with a screen, camera, microphone, and speaker (smartphone, tablet, or computer); and
* Have a reasonable self-assessment ability to use the internet (through a 4-item scale from poor, fair, good to excellent).

Exclusion Criteria:

* History of traumatic injury.
* Previous surgery related to the lumbar spine.
* Undergoing cancer treatment.
* Presenting with any inflammatory rheumatological condition.
* Decompensated cardiovascular disorders.
* Presence of comorbidity or condition that may hinder active participation in the prescribed exercises to be performed at home.
* Severe psychological disorders.
* Pregnant individuals.
* Awaiting surgical procedure.
* Having undergone intervention including exercise or physiotherapeutic treatment in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | The participants' pain intensity will be evaluated at baseline (T0), after 12 sessions (T1), at 3 months (T2), and at 6 months (T3).
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS). It is an 11-point scale ranging from 0 to 10, with zero indicating no pain and 10 indicating the most unbearable pain experienced by the participant. The subject will be asked about the presence of pain specifically localized to the lumbar region. Additionally, the frequency (every day, more than 15 days per month, between 8 and 15 days per month, between 1 and 7 days per month, or between 4 and 11 crises per year) and duration of symptoms (less than 2 years, 2 to 5 years, 6 to 10 years, more than 10 years) will be queried. The following definition of LBP will be utilized: "pain in the area between the 12th rib and the gluteal fold with or without leg pain.

SECONDARY OUTCOMES:
Functional disability | The participants' functional disability will be evaluated at baseline (T0), after 12 sessions (T1), at 3 months (T2), and at 6 months (T3).
  The Roland-Morris Disability Questionnaire (RMDQ) will be used. This questionnaire assesses the impact of low back pain on work and daily life activities due to symptoms, and it is better recommended for a population with low functional disability. The instrument has been validated for Brazilian Portuguese, is quick and easy to administer, with an average response time of five minutes. Scores are obtained by summing the items, which range from zero (no disability) to 24 (severe disability). Scores higher than 14 indicate physical disability. The minimum clinically important difference is 5 points.
Quality of life Impact | The participants' quality of life will be evaluated at baseline (T0), after 12 sessions (T1), at 3 months (T2), and at 6 months (T3).
  To assess quality of life, the 12-Item Short-Form Health Survey (SF-12) will be used as a quicker alternative to the 36-Item Health Survey. Comprising twelve items derived from the SF-36, the SF-12 assesses eight different dimensions influencing quality of life, considering the individual's perception of their health over the past four weeks. Each item has a set of responses distributed on a Likert-type scale, evaluating the following dimensions: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Through the instrument's own algorithm, two scores can be measured: the physical component summary (PCS) and the mental component summary (MCS). In both, scores range from 0 to 100 points, with higher scores associated with better quality of life. Psychometric properties of the instrument have also been evaluated.
State-Trait Anxiety | The participants' State-Trait Anxiety will be evaluated at baseline (T0), after 12 sessions (T1), at 3 months (T2), and at 6 months (T3).
  For anxiety assessment, the State-Trait Anxiety Inventory (STAI) will be used, which has been translated and adapted for use in Brazil. The scale consists of 2 self-report scales that assess state and trait anxiety. The scale comprises 20 items scored from 1 to 4 each, resulting in a total score ranging from 20 to 80 points. For each question, the corresponding score is assigned, but for positively framed questions, the score is reversed. Scores > 42 tend to indicate anxiety, while scores < 38 tend to indicate depression. The STAI Manual suggests using the title "Self-Assessment Questionnaire" instead of the term Anxiety.
Fear Avoidance Beliefs | The participants' fear avoidance beliefs will be evaluated at baseline (T0), after 12 sessions (T1), at 3 months (T2), and at 6 months (T3).
  The Fear Avoidance Beliefs Questionnaire (FABQ), translated into Brazilian Portuguese, contains two sub-scales that are evaluated separately: fear-avoidance beliefs related to work (FABQ-work) and physical activity (FABQ-physical). Fear avoidance related to physical activity will be considered present (score ≥15) or absent (<15), while fear avoidance related to work will be considered present if the FABQ-work score is ≥ 34.

OTHER OUTCOMES:
Sociodemographic and clinics characteristics | The Sociodemographic and clinics characteristics will be evaluated at baseline (T0).
  Sociodemographic characteristics (gender, age, marital status, self-declared race), socioeconomic factors (years of education and individual income), main occupational activity they have performed throughout their lives, and whether they are still engaged in it at the time of the research, according to the Brazilian Classification of Occupations. Clinical characteristics will include anthropometric variables: self-reported weight and height for subsequent calculation of Body Mass Index, stratified according to age groups as recommended by the World Health Organization, alcohol and tobacco consumption, self-reported diseases, and behavioral variables such as level of physical activity assessed by the International Physical Activity Questionnaire. Additionally, participants will be asked about medication consumption, dosages, seeking healthcare professionals for LBP treatment.
Perception of discrimination | The Perception of Discrimination will be evaluated at 6 months (T3).
  For the assessment of Perception of Discrimination, the adaptation of the "Everyday Discrimination to the context of healthcare utilization" scale and adapted for the healthcare context will be used. It consists of 7 qualitative statements about the experience during the search for and treatment of the health condition, in this case, for LBP, and the higher the score, the more present the perception of discrimination.

CONTACTS AND LOCATIONS:
Overall Officials: Ingred Merllin B de Souza, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- Dept. Physical Therapy, Audiology and Speech Therapy at Medical School, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT06443229/SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT06443229/ICF_001.pdf